CLINICAL TRIAL: NCT04444219
Title: Postprandial Glucose, Insulin Responses and Appetite Hormones to Dried Mushrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assosiate Professor in Foods and Human Nutrition, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Nutritious_Mushrooms_Postprand
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Breakfast

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breakfast meal_1 (Other): 100 g white bread, 40 g yellow cheese and Κing Oyster mushrooms (test meal)
  Interventions: Other: Breakfast meals
- Breakfast meal_2 (Other): 100 g white bread, 40 g yellow cheese and 6-7 cherry tomatoes (control meal)
  Interventions: Other: Breakfast meals

INTERVENTIONS:
Other: Breakfast meals — Fifteen volunteers will undergo a medical and dietary assessment and their health status will be evaluated through a complete blood count. Then, they will come after overnight fasting and will consume one of two breakfast meals, including 114g bread, 40g cheese and 15g dry mushrooms (meal 1) or 114g bread, 40g cheese and 200g tomatoes (meal 2). Blood samples will be obtained on timepoints 0h, 30min, 1h, 1,5h, 2h, 2,5h and 3h after breakfast intake. Two weeks later, the same volunteers will consume the other breakfast meal.

SUMMARY:
Obesity, characterized by an increase in body weight that results in excessive fat accumulation, is a global health problem. Recently, it has also been shown that obesity is associated with low-grade chronic systemic inflammation in adipose tissue. This condition is mediated by activation of the innate immune system in adipose tissue that promotes inflammation and oxidative stress and triggers a systemic acute-phase response.

Previous research points towards the potential of phytochemicals in food as part of nutritional strategies for the prevention of obesity and associated inflammation, as well as, increase in insulin sensitivity in diabetic patients.

The last decade, mushrooms have attracted the research interest as functional foods rich in beta-glucan with desirable health benefits in several metabolic disorders without the side effects of pharmacological treatment. Edible mushrooms are highly nutritious and exhibit beneficial effects on several inflammatory diseases such as cancer, heart disease, diabetes,, high blood pressure.

However, the postprandial effect of mushrooms in human biological samples is still undetermined. To this end, the current study aims to investigate if there is any effect at postprandial glucose, insulin responses and appetite hormones. Fifteen apparently men and women with Metabolic Syndrome, aged 18-65 years old, will be enrolled based on certain inclusion and exclusion criteria.

After enrollment, the volunteers will undergo a medical and dietary assessment and their health status will be evaluated through a complete blood count. On the day of the experiment and after overnight fasting, the volunteers will consume one of two breakfast meal, including 114g bread, 40g cheese and 15g dry mushrooms (meal 1) or 114g bread, 40g cheese and 200g tomatoes (meal 2). Blood samples will be obtained on timepoints 0h, 30min, 1h, 1,5h, 2h, 2,5h and 3h after breakfast intake. Two weeks later, the same volunteers will consume the other breakfast meal.

After collection, the glucose and insulin values will be identified in plasma samples. Additionally, some appetite hormones will be measureD in serum samples.

ELIGIBILITY:
Inclusion Criteria:

18 years < Age < 75 years BMI > 25 kg/ m2 Metabolic Syndrome

Exclusion Criteria:

Hepatotoxic Medication Diabetes Mellitus Dysthyroidism, hypopituitarism, Cushing syndrome / disease Pregnancy, lactation Psychiatric or mental disorder Any use of antioxidant-phytochemical rich supplement, vitamin D supplement, nti-, pre- or pro-biotics within 3 months pre-intervention

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Difference of Glucose levels | 1 month
  Difference of Glucose levels after consuming the two meals
Difference of Insulin levels | 1 month
  Difference of insulin levels after consuming the two meals
Difference of appetite hormones levels | 1 month
  Difference of appetite hormones levels after consuming the two meals

CONTACTS AND LOCATIONS:
Locations (1):
- Andriana Kaliora, Athens, Greece

REFERENCES:
- [Background] Marseglia L, Manti S, D'Angelo G, Nicotera A, Parisi E, Di Rosa G, Gitto E, Arrigo T. Oxidative stress in obesity: a critical component in human diseases. Int J Mol Sci. 2014 Dec 26;16(1):378-400. doi: 10.3390/ijms16010378. PMID 25548896
- [Background] Cardwell G, Bornman JF, James AP, Black LJ. A Review of Mushrooms as a Potential Source of Dietary Vitamin D. Nutrients. 2018 Oct 13;10(10):1498. doi: 10.3390/nu10101498. PMID 30322118
- [Background] Abdali D, Samson SE, Grover AK. How effective are antioxidant supplements in obesity and diabetes? Med Princ Pract. 2015;24(3):201-15. doi: 10.1159/000375305. Epub 2015 Mar 14. PMID 25791371
- [Background] El Khoury D, Cuda C, Luhovyy BL, Anderson GH. Beta glucan: health benefits in obesity and metabolic syndrome. J Nutr Metab. 2012;2012:851362. doi: 10.1155/2012/851362. Epub 2011 Dec 11. PMID 22187640
- [Background] Ganesan K, Xu B. Anti-Obesity Effects of Medicinal and Edible Mushrooms. Molecules. 2018 Nov 5;23(11):2880. doi: 10.3390/molecules23112880. PMID 30400600